CLINICAL TRIAL: NCT06587165
Title: A Pilot Study for Quantifying New Heart Muscle Cells
Brief Title: Quantifying New Heart Muscle Cells
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); California Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-03027194; 7R01HL151386-05 (NIH)
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Tetralogy of Fallot With Pulmonary Stenosis; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- N15-thymidine (Experimental): Study participants will receive thymidine preparations for pre-defined blocks of time prior to the scheduled routine resection of myocardium.
  Interventions: Other: N15-thymidine

INTERVENTIONS:
Other: N15-thymidine — 50mg/kg (oral administration)

SUMMARY:
Regenerative therapies could provide new ways of treating heart failure. Unlike many organs in the human body, such as the skin and the GI tract, the ability to regenerate heart muscle decreases after birth, but the precise timing of this decrease and how this decrease is altered in heart disease are uncertain. The investigators will use an innovative approach to quantify cellular heart regeneration in pediatric patients, an appropriate population for determining this decline as well as the potential for reactivating heart muscle regeneration.

The study has now been registered on ClinicalTrials.gov, despite its initiation on July 23, 2015, as registration was not mandated at the original study site, the University of Pittsburgh Medical Center. However, following the transfer of the study to Weill Cornell Medicine, adherence to institutional requirements necessitated its registration on ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Patients at 30 days of age to 1 year of age undergoing scheduled elective cardiac surgery will be eligible for study inclusion.
* The investigators will recruit patients at 30 days of age to 1 year of age with those types of heart disease whose surgical approach has a high probability of myocardial resection.
* Diagnosis of ToF/PS or other types of heart disease that have a high likelihood of requiring surgery that involves routine resection of myocardium that becomes available for research

Exclusion Criteria:

* Patients with low chance of having resection of myocardium as part of their surgical care.

Ages: 30 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-07-23 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of labeled cardiomyocytes for each patient | 6 months
  The investigators will use, multi-isotope imaging mass spectrometry (MIMS) to quantify the generation of new cardiomyocytes by examining myocardial samples that are routinely resected and discarded during cardiac surgery. Investigators will then calculate the percentage of labeled, i.e. newly generated, cardiomyocytes, for each patient. The data from the analysis of myocardial samples will be the test results. Investigators will first compare these results with technical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Kuhn, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No